CLINICAL TRIAL: NCT02454712
Title: A Phase 1, Single-Center, Dose-Escalation Study to Determine the Safety and Pharmacokinetics of a Single Oral Dose of PF614 in Healthy Subjects Compared to OxyContin®
Brief Title: Study of PF614 Compared to OxyContin® in Healthy Volunteers (PF614-101)
Acronym: SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ensysce Biosciences (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PF614-101
Record Dates: First submitted 2015-05-12; First posted 2015-05-27 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Prodrug; PF614; oxycodone extended-release; oral
MeSH Terms: interventions — Oxycodone; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PF614 (Experimental): PF614 is the drug under evaluation. Doses may range from 15 mg to 640 mg. N=6 subjects per cohort. For Cohort 7, N=16 subjects in crossover study ± naltrexone.
  Interventions: Drug: PF614; Drug: Naltrexone Hydrochloride
- Oxycodone extended-release (OxyContin) (Active Comparator): Initial dose (Cohort 1) will be 10 mg. Subsequent doses will be 10, 20, 40, or 80 mg. N=2 subjects per cohort. Active comparator will not be used in Cohort 7.
  Interventions: Drug: Oxycodone extended-release; Drug: Naltrexone Hydrochloride

INTERVENTIONS:
Drug: PF614 — PF614 is an oxycodone prodrug
  Other Names: PRF06104
  Arms: PF614
Drug: Oxycodone extended-release — Oxycodone extended-release is the comparator drug
  Other Names: OxyContin
  Arms: Oxycodone extended-release (OxyContin)
Drug: Naltrexone Hydrochloride — Naltrexone HCl tablets, 50 mg, will be used to block high dose opioid effects in healthy volunteers
  Other Names: ReVia

SUMMARY:
PF614 is an oxycodone prodrug that is designed for extended-release of oxycodone comparable to OxyContin. This Single Ascending Dose (SAD) study is designed to assess the safety and pharmacokinetics (PK) of PF614 in comparison to standard doses of OxyContin.

DETAILED DESCRIPTION:
This will be a Phase 1 randomized, single-center, SAD study in 6 cohorts of 8 healthy male and/or female subjects each (Cohorts 1-6) plus 16 enrolled healthy male and/or female subjects (Cohort 7). The study will evaluate the safety and PK of PF614 and the PK of oxycodone at doses sufficient to characterize the extent to which plasma oxycodone is produced and maintained following oral ingestion of PF614. The PK of the prodrug fragments will also be evaluated. There will be a parallel study arm in each cohort dosed that will use oral OxyContin® as an active comparator. Subjects will receive PF614 (n=6) or OxyContin as comparator (n=2) orally in the fasted state. In addition, all subjects starting with Cohort 1C will receive naltrexone at 14 hours pre-dose, 2 hours pre-dose and 10 hours post dose to block the effects of oxycodone. The starting dose for administration of PF614 will be 15 mg. The lowest available dose of OxyContin, 10 mg, will be used as the comparator in the first cohort. PK assessments will be conducted after each cohort to compare the oxycodone area under curve (AUC) of PF614 and OxyContin to determine the most appropriate dose for the subsequent cohorts. In Cohort 6 (fed subjects), all subjects (n=8) will receive the same PF614 and naltrexone doses as administered in Cohort 5 to evaluate the PK and safety of PF614 in fed vs. fasted state. Subjects in Cohort 6 will receive a Food and Drug Administration-defined high-fat, high-calorie breakfast 30 minutes prior to study drug administration. In Cohort 7, treatments will be administered in a cross-over study design across 2 periods. All subjects (n=16 enrolled; estimated n=12 completers) will receive the same PF614 dose as administered in Cohort 1 (15 mg) with and without naltrexone to evaluate the potential effect of naltrexone on the plasma PK of PF614 and oxycodone. Cohort 7, Period 1 subjects may return for their cross-over treatments in Period 2 after a minimum of 12 days after receiving their initial Cohort 7 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ages 18-50 years (inclusive) in good general health;
2. Body mass index (BMI) between 18.0 and 32.0 kg/m2 (inclusive);
3. Minimum weight of 50.0 kg, inclusive;
4. Subjects must have a negative screen for drugs of abuse, cotinine, alcohol, hepatitis B-surface antigen, hepatitis C antibody and antibodies against HIV 1 and 2;
5. Female subjects must have a negative serum pregnancy test at screening and a negative pregnancy test on Day -1;
6. Females of childbearing potential and males and their female partner(s) of childbearing potential must agree to use 2 forms of contraception, 1 of which must be a barrier method, during the study and for 90 days after the last drug administration. Acceptable barrier forms of contraception are condom and diaphragm. Acceptable nonbarrier forms of contraception for this study are a nonhormonal intrauterine device (IUD), oral contraceptives and/or spermicide;
7. Male subjects must agree not to donate sperm throughout the study and for 90 days after the last study drug administration;
8. Subjects must have normal or no evidence of clinically significant findings in physical examination and 12-lead electrocardiogram (ECG) according to the Investigator, and normal vital signs (respiratory rate between 10 and 18 breaths per minute, blood pressure between 100-139/50-89 mmHg, heart rate between 40-100 beats per minute, temperature between 96.44°F and 100.04°F (between 35.8°C and 37.8°C), and oxygen saturation (SpO2) > 97% in the absence of supplemental oxygen;
9. Clinical laboratory values must be within the normal limits as defined by the clinical laboratory, unless the Investigator decides that out-of-range values are not clinically significant;
10. Subjects must be able to provide meaningful written informed consent;
11. Subjects must be willing and able to follow study instructions and be likely to complete all study requirements.

Exclusion Criteria:

1. History of allergy or sensitivity to oxycodone, OxyContin, any other opiate, naltrexone, or naloxone;
2. History of loud snoring or sleep apnea;
3. History of medical problems encountered with opioid therapy;
4. Urinary cotinine levels indicative of smoking or history of regular use of tobacco-containing or nicotine-containing products within 2 months prior to screening;
5. History of alcoholism or drug abuse (prescription or illicit drugs) according to Diagnostic and Statistical Manual IV-Text Revision (DSM IV-TR) criteria;
6. Use of prescription medications within 14 days of study drug administration, except for contraceptive medications used by female subjects; use of over-the-counter (OTC) medications within 7 days prior to study drug administration;
7. Use of any opioid within 30 days prior to screening;
8. Donation of blood within 60 days prior to screening;
9. Donation of plasma, platelets, or white blood cells within 7 days prior to dosing;
10. Acute illness (eg, gastrointestinal illness, infection such as influenza, upper respiratory tract infection, or known inflammatory process) within 7 days of dosing
11. History of gastrointestinal disturbance requiring frequent use of antacid;
12. History of clinically significant gastrointestinal disease and/or surgery which would result in the subject's inability to absorb or metabolize the study drug (eg, gastrectomy, gastric bypass, cholecystectomy);
13. Anticipated need for surgery or hospitalization during the study or follow-up period;
14. Dosing with an investigational drug or participation in an investigation device study within 30 days or 5 half-lives of first dose of the study drug;
15. Women who are lactating;
16. Any other condition, that, in the Investigator's opinion, (i) puts the subject at increased risk, (ii) could confound the study results (iii) may interfere significantly with the subject's participation in the study or (IV) has the potential to limit the subject's ability to complete the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Safety | 30 days
  Adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours post dose
  Peak plasma concentrations of oxycodone derived from PF614 and OxyContin
Pharmacokinetics (Tmax) | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours post dose
  Time to peak plasma concentrations of oxycodone derived from PF614 and OxyContin
Pharmacokinetics (AUC) | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours post dose
  Area under the plasma concentration vs. time curve (AUC) for oxycodone derived from PF614 and OxyContin
Dose Selection (Identify doses of PF614 with pharmacokinetics comparable to OxyContin) | 4 days
  Identify doses of PF614 with pharmacokinetics comparable to OxyContin
Prodrug Fragments (plasma concentration) | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours post dose
  Evaluate appearance and plasma concentrations of metabolic fragments derived from PF614
Pharmacokinetics (Cmax) in fed vs. fasted state | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours post dose
  Peak plasma concentrations of oxycodone derived from PF614
Pharmacokinetics (Tmax) in fed vs. fasted state | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours post dose
  Time to peak plasma concentrations of oxycodone derived from PF614
Pharmacokinetics (AUC) in fed vs. fasted state | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours post dose
  Area under the plasma concentration vs. time curve (AUC) for oxycodone derived from PF614
Effect of naltrexone on PF614 and oxycodone plasma PK in a crossover design | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours post dose
  Cmax and AUC of plasma oxycodone

CONTACTS AND LOCATIONS:
Overall Officials: William K Schmidt, PhD, Study Director — Ensysce Biosciences
Locations (1):
- PRA Health Sciences - Early Development Services, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt WK, Dickerson DS, Fisher DM, Kirkpatrick DL. First-in-human pharmacokinetics & safety study of PF614: orally activated oxycodone prodrug. Anesth Analg. 2017;124(5):752-753.
- [Background] Kirkpatrick DL, Evans C, Pestano LA, Millard J, Johnston M, Mick E, Schmidt WK. Clinical evaluation of PF614, a novel TAAP prodrug of oxycodone, versus OxyContin in a multi-ascending dose study with a bioequivalence arm in healthy volunteers. Clin Transl Sci. 2024 Mar;17(3):e13765. doi: 10.1111/cts.13765. PMID 38511523